CLINICAL TRIAL: NCT02631434
Title: Comparison Between Sit-to-stand Test and Six-minute Walk Test in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STSTCOPD
Record Dates: First submitted 2015-11-25; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sit-to-stand (Experimental): To perform a sit-to-stand test
  Interventions: Procedure: sit-to-stand test
- six minute walking test (Active Comparator): To perform a six minutes walking test
  Interventions: Procedure: six-minutes walking test

INTERVENTIONS:
Procedure: sit-to-stand test
  Arms: sit-to-stand
Procedure: six-minutes walking test
  Arms: six minute walking test

SUMMARY:
Comparison between sit-to-stand test and six minutes walking test in chronic obstructive pulmonary disease patients

ELIGIBILITY:
Inclusion Criteria:

* clinically stable for a minimum of 4 weeks
* no recent infectious exacerbations

Exclusion Criteria:

* musculoskeletal or joint disorders
* contra-indications to perform exercises

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
number of sit-to-stand movement | 1 minute
walked distance | 6 minutes

SECONDARY OUTCOMES:
heart rate | 6 minutes
fraction of oxygen-saturated hemoglobin measured by pulsed oximeter | 6 minutes
breathlessness measured by visual analogic scale | 6 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique universitaire Saint-Luc, Brussels, Belgium